CLINICAL TRIAL: NCT06747377
Title: Evaluation of Left Ventricular Function After Treatment of Diabetic Foot Ulcers Using Longitudinal Strain Echocardiography
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amal Refaie Ahmed Ali, resident doctor Assiut University hospital, Assiut University
Other Study IDs: LVF strain echocardiography
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Foot Ulcers (DFU)
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- diabetic foot ulcer: Diabetic Patients with DFU, who were diagnosed by a vascular surgeon based on Diabetic Foot Study Group guidelines.

SUMMARY:
Early detection of heart failure as a macrovascular complication of DM offers the best chance of cure in these patients. Nowadays, the most common method for detecting heart failure is measuring left ventricle ejection fraction (LV-EF), by echocardiography. Despite the easy application of LV-EF, it remains normal in early stages of cardiac disease and it's considered as heart failure with preserved LVEF (HFpEF). We hope that, Strain monitoring as a new method enables us to detect the early minimal changes in myocardium.

The aim of study evaluate the effect of treatment of diabetic foot ulcers in improving heart function by strain echocardiography than conventional transthoracic echocardiography in Assiut university hospital.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a chronic, metabolic disease with hyperglycemia that occurs as a result of deficiency or resistance of insulin hormone secreted from the pancreas. Diabetic foot ulcer (DFU)is a frequent macrovascular complication has a high incidence and mortality rate. According to research statistics, the mortality rate of patients with foot ulcers after 5 years is 2.5 times higher than that of patients without such ulcers. Heart failure develops in diabetic patients over twice higher than non-diabetics both directly, by impairing cardiac function, and indirectly, through associated diseases such as hypertension, coronary disease, renal dysfunction, obesity, and other metabolic disorders.

Based on a recent study, DFU treatment improves cardiac function assessed by strain measurements . At present, few data is available about the ability of strain echocardiography in prediction of systolic dysfunction in DFU, and the possible effect of the treatment of these patients on their cardiac function. So, we decided to evaluate the effect of treatment of diabetic foot ulcers in improving heart function by this new method-strain echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic Patients with DFU, who were diagnosed by a vascular surgeon based on Diabetic Foot Study Group guidelines.
* Diabetic Patients were who used anti-diabetic oral medication, insulin or who had fasting blood glucose (FBS) ≥ 126 mg/dl for at least two times at age group 18 to 50 years at Assiut university hospital

Exclusion Criteria:

* Patients with acute or advanced stage of renal, hepatic or pulmonary diseases, acute coronary syndrome, known coronary artery disease ,infectious disease in the last two weeks, coagulopathy, history of a hemorrhagic stroke, severe valvular disease , heart failure (EF<45%).
* at age group below 18 or above 50 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Group guidelines.
  -Diabetic Patients were who used anti-diabetic oral medication, insulin or who had fasting blood glucose (FBS) ≥ 126 mg/dl for at least two times at age group 18 to 50 years at Assiut university hospital
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
cure rate | baseline
  cure rate after Diabetic foot ulcers treatment in patients who suffer from this condition can lead to an improvement in cardiac function,

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jin Y, Meng M, Zhang Y, Mo L, Gao H, Liu Y, Wu J, Yang P, Zhang Z, Jia F, Zhao Y, Huang Y. Comparative study on the efficacy of PRP gel and UC-MSCs gel as adjuvant therapies in the treatment of DFU wounds. Skin Res Technol. 2024 Jan;30(1):e13549. doi: 10.1111/srt.13549. PMID 38174781